CLINICAL TRIAL: NCT05153252
Title: Does When You Exercise Matter? A Randomized Trial Comparing the Effect of Morning Versus Evening Aerobic Exercise on Weight Loss and Compensatory Behaviors
Brief Title: Timing Intervention of Morning Versus Evening Exercise
Acronym: TIMEX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-3094; 1R01DK126814-01A1 (NIH)
Record Dates: First submitted 2021-11-23; First posted 2021-12-10 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Overweight and Obesity
Keywords: Overweight; Obesity; Exercise
MeSH Terms: conditions — Overweight; Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morning Exercise (AM) (Experimental): Participants in this group will be prescribed morning aerobic exercise.
  Interventions: Behavioral: Morning Exercise
- Evening Exercise (PM) (Experimental): Participants in this group will be prescribed evening aerobic exercise.
  Interventions: Behavioral: Evening Exercise

INTERVENTIONS:
Behavioral: Morning Exercise — Morning Exercise will be instructed to perform 2000 kcal/wk of moderate to vigorous intensity aerobic exercise between the hours of 6 and 10 AM.
  Other Names: AM Exercise; AM-EX
  Arms: Morning Exercise (AM)
Behavioral: Evening Exercise — PM will be instructed to perform 2000 kcal/wk of moderate to vigorous intensity aerobic exercise between the hours of 3 and 7 PM.
  Other Names: PM Exercise; PM-EX
  Arms: Evening Exercise (PM)

SUMMARY:
The investigators are doing this study to learn more about how exercising at different times of the day (morning versus evening) affects body weight, sleep, eating patterns, and other factors.

DETAILED DESCRIPTION:
Does the time of day that exercise is performed matter for weight loss? The objective of this proposal is to examine the impact of an equivalent dose of morning vs. evening aerobic exercise on change in body weight, energy intake (EI) and components of energy expenditure (EE) in adults with overweight or obesity. Nearly two-thirds of US adults who attempt to lose weight report engaging in exercise as a primary strategy for weight loss. However, weight loss from exercise alone is often substantially less than predicted based on calories burned in exercise. This is due to compensatory changes that occur in response to exercise initiation (e.g. increases in EI and decreases in non-exercise EE) that limit the energy deficit produced by exercise. Thus, strategies that reduce the compensatory response to exercise could enhance the weight loss efficacy of exercise. It is possible that exercise time of day could impact compensatory behaviors and weight loss, however, there have been no adequately powered, prospective, randomized studies comparing weight loss induced by morning vs. evening exercise. The study design is a 7-month supervised trial in which adults with overweight or obesity will be randomized to supervised aerobic exercise (2000 kcal/wk) performed either in the morning (AM-Ex, 6-10 AM) or the evening (PM-Ex, 3-7 PM). The supervised exercise phase will be followed by a 6-month maintenance phase during which participants continue to exercise at the target of 2000 kcal/week during the randomized AM or PM exercise windows, but exercise is no longer supervised. Aim 1 will compare the effects of AM-Ex vs. PM-Ex on changes in body weight and body composition with the primary study outcome of weight change at 7-months. Aim 2 will compare the effects of AM-Ex vs PM-Ex on changes in EI and appetite. Aim 3 will compare the effects of AM-Ex vs PM-Ex on changes in EE, non-exercise physical activity and sedentary time. Exploratory Aim 4 will compare the effects of AM-Ex vs PM-Ex on changes in meal and sleep timing. This approach is rigorous and innovative as the exercise energy deficit will be matched between groups, exercise will be prescribed based on EE, and free-living total daily energy expenditure (TDEE) and EI will be assessed objectively (using doubly-labeled water). This study is significant as it could provide important insight on how the timing of exercise impacts weight loss and compensatory behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Female or Male
* Age 18-55 years
* Body Mass Index 25-40 kg/m2
* Physically inactive: defined as self-reporting <150 minutes per week of physical activity at moderate intensity or greater on a regular basis over the past 3 months.
* No self-report of acute or chronic disease (cardiovascular disease (CVD), diabetes, gastrointestinal disorders and orthopedic problems in particular)
* No plans to relocate within the next 15 months.
* No plans for extended travel (> 2 weeks) within the next 13 months
* Live or work within 30 minutes of the Anschutz Health & Wellness Center (AHWC) (exceptions may be made at the discretion of the Study PI on a case-by-case basis for highly motivated subjects).
* Capable and willing to give informed consent, understand exclusion criteria, accept the randomized group assignment, and complete outcome measures.
* No contraindications to exercise or limitations on ability to be physically active.
* Willing to be randomized to either AM or PM exercise and complete 4 exercise sessions per week.
* Own a smart phone and willing to download and use text messaging for meal intake and other related assessments.
* Willing and able to wear activity/sleep monitor for 7-14 consecutive days.
* Willing not to enroll in any other formal weight loss or physical activity programs over the next 13 months.
* Fully vaccinated, or willing to be fully vaccinated, against COVID-19 prior to study enrollment (fully vaccinated is defined as at least 2 weeks post final vaccine dose).
* Have a primary care physician (or are willing to establish care with a primary care physician prior to study enrollment) to address medical issues which may arise during screening or study procedures/interventions.
* For Females

  * Not currently pregnant or lactating
  * Not pregnant within the past 6 months
  * Not planning to become pregnant in the next 15 months; sexually active women of childbearing potential may be enrolled if they have had a tubal ligation or use a reliable means of contraception

Exclusion Criteria:

* Diastolic blood pressure > 100 mm HG or systolic blood pressure > 160 mm HG.
* Resting heart rate >100
* Diabetes (fasting glucose ≥126 mg/dL or Hemoglobin A1C ≥6.5%)
* Undiagnosed hypo- or hyper-thyroidism (Thyroid Stimulating Hormone (TSH) outside of the normal range) or history of uncontrolled thyroid disorder. History of thyroid disease or current thyroid disease treated with a stable medication regimen for at least 6 months is acceptable.
* Hematocrit, white blood cell count or platelets significantly outside the normal reference range.
* Clinically significant abnormalities in hematocrit, white blood cell count or platelets.
* Triglycerides > 400 mg/dL
* (Low Density Lipids) LDL cholesterol >200 mg/dL
* Abnormal resting electrocardiogram (ECG): serious arrhythmias, including multifocal premature ventricular contractions (PVC's), frequent PVC's (defined as 10 or more per min), ventricular tachycardia (defined as runs of 3 or more successive PVC's), or sustained atrial tachyarrhythmia; 2nd or 3rd degree A-V block, QTc interval > 480 msec or other significant conduction defects.
* Presence or history of any metabolic or chronic health problems which would affect appetite, food intake, energy metabolism, or ability to optimally participate in the exercise component including: CVD, peripheral vascular disease, cerebrovascular disease, significant cardiac arrhythmias or cardiac valve disease, diabetes, uncontrolled hyper- or hypothyroidism, uncontrolled hypertension, cancer (within the last 5 years, except skin cancer or other cancers considered cured with excellent prognosis), HIV infection, significant gastrointestinal disorders (described below), significant pulmonary disorders (described below), significant renal, musculoskeletal, neurologic, hematologic, or psychiatric disease.
* Significant gastrointestinal disorders including: Crohn's disease, Ulcerative Colitis, chronic diarrhea, or active gallbladder disease.
* Significant pulmonary disorders including: chronic obstructive pulmonary disease (COPD), interstitial lung disease, cystic fibrosis, or uncontrolled asthma.
* Symptoms suggestive of CVD: chest pain, shortness of breath at rest or with mild exertion, syncope.
* Regular use of prescription or over-the-counter medications known to significantly impact appetite, weight, sleep, or energy metabolism (e.g., appetite suppressants, lithium, stimulants, anti-psychotics, tricyclic antidepressants)
* Use of medications that would impact ability to achieve age-predicted maximum heart rate (e.g. beta blockers, cardio-selective calcium channel blockers).
* Regular use of systemic steroids (other than Oral Contraceptive Pills)
* Regular use of obesity pharmacotherapeutic agents within the last 6 months.
* Previous obesity treatment with surgery or weight loss device, except: (1) liposuction and/or abdominoplasty if performed > 1 year before screening, (2) lap banding if the band has been removed > 1 year before screening, (3) intragastric balloon if the balloon has been removed > 1 year before screening (4) duodenal-jejunal bypass sleeve, if the sleeve has been removed > 1 year before screening or 5) AspireAssist or other endoscopically placed weight loss device if the device has been removed > 1 year before screening.
* Current alcohol or substance abuse
* Nicotine use (past 6 months)
* History of clinically diagnosed eating disorders including anorexia nervosa, bulimia, binge eating disorder. Score >20 on the Eating Attitudes Test (EATS-26) or pattern of response on the Questionnaire on Eating and Weight Patterns (QEWP-5) suggestive of possible binge eating disorder or bulimia will require further assessment by the Study MD to determine if it is appropriate for the subject to participate in the study.
* Current severe depression or history of severe depression within the previous year, based on Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR) criteria for Major Depressive Episode. Score > 18 on Beck Depression Inventory (BDI) will require further assessment by the Study MD to determine if it is appropriate for the subject to participate in the study.
* History of other significant psychiatric illness (e.g. psychosis, schizophrenia, mania, bipolar disorder) which in the opinion of the Study MD would interfere with ability to adhere to dietary or exercise interventions.
* Night-time shiftwork, rotating work, irregular sleep/wake patterns or other scheduling constraints which may hinder ability to consistently exercise at specific times of the day.
* Urinary incontinence or retention (as per PI discretion based on whether degree of incontinence/retention may impact doubly labeled water measures).
* Weight loss >5% in past 3 months.
* Weight gain >10% in past 3 months requires assessment by PI to determine reason for weight gain and if it is appropriate for the subject to participate in the study.
* Weight loss of >50 lbs in past 3 years for any reason except post-partum weight loss requires assessment by PI to determine reason for weight gain and if it is appropriate for the subject to participate in the study.
* Currently participating in or planning to participate in any formal weight loss, dietary modification, or physical activity/exercise programs or clinical trials.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2021-12-07 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Weight Change (kg) | Baseline (0) - 13 Months
  Body weight will be measured using a digital scale at baseline, 3.5, 7, and 13 months. The primary outcome will be change in weight from baseline to 7 months.

SECONDARY OUTCOMES:
Fat Mass | Baseline (0) - 13 Months
  Fat mass will assessed using Dual-Energy X-Ray Absorptiometry (DXA) at baseline, 7, and 13 months.
Lean Mass | Baseline (0) - 13 Months
  Lean Mass will assessed using Dual-Energy X-Ray Absorptiometry (DXA) at baseline, 7, and 13 months.
Energy Intake | Baseline (0) - 7 Months
  Energy Intake (EI) will be assessed using the Doubly Labeled Water (DLW) Intake-Balance Method at baseline and 7
Total Daily Energy Expenditure | Baseline (0) - 7 Months
  Total Daily Energy Expenditure (TDEE) will be assessed using doubly labeled water (DLW) at baseline and 7 months
Hunger and Satiety | Baseline (0) - 13 Months
  Assessed with visual analog scale (0-100 range). Higher scores indicate higher levels of hunger (worse outcome) and satiety (better outcome). Measured at baseline, 3.5, 7, and 13 months
Food Cravings | Baseline (0) - 13 Months
  Assessed with 2 questionnaires at baseline, 3.5, 7, and 13 months: Food Cravings Questionnaire Trait-reduced (FCQ-T-r) and and FCI-II. Higher scores indicate greater cravings (worse outcome). Food Cravings Questionnaire-Trait-reduced (FCQ-T-r) is a Likert Scale using scoring associated with it Strongly disagree = 1, Disagree = 2, Neither agree nor disagree = 3, Agree= 4, Strongly agree = 5. The FCI-II is scored on a Likert scale from 1-5, with 1 being "Never," 5 being "Always/Almost every day." It has 4 subscales: High Fats, Sweets, Carbohydrates/Starches, and Fast-Food Fats. The score for each subscale is obtained by averaging the responses to the items listed for the subscale. The total score is obtained by averaging the responses to all 28 items.
Aspects of Eating Behavior | Baseline (0) - 13 Months
  Measured via Three-Factor Eating Questionnaire at baseline, 3.5, 7, and 13 months. This assessment is designed to measure 3 dimensions of human eating behavior: cognitive restraint of eating (Factor I - 20 items), disinhibition (Factor II - 16 items), and hunger (Factor III - 15 items). The minimum score for factors I-II-III is therefore 0-0-0, and maximum possible score is 20-16-15. Part I includes items 1-36 and are rated either 1-True or 0-False. Part II includes items 37-51 and is rated on a 4-point scale with the exception of item 50, which is rated on a 6-point scale.
Non-Exercise Physical Activity (NEPA) | Baseline (0) - 13 Months
  NEPA will be measured with the ActivPAL device at baseline, 3.5, 7, and 13 months
Sedentary Time | Baseline (0) - 13 Months
  Sedentary Time will be measured with the ActivPAL device at baseline, 3.5, 7, and 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Vicki Catenacci, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-08-03): https://cdn.clinicaltrials.gov/large-docs/52/NCT05153252/ICF_000.pdf